CLINICAL TRIAL: NCT01230229
Title: Primary Stenting vs Conservative Treatment in Claudicants - a Study on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Anders Gottsater, MD, PhD, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SFA stenting and QoL
Record Dates: First submitted 2010-10-28; First posted 2010-10-29 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Stable Claudication (Fontaine IIa and IIb); Superficial Femoral Artery Disease; Best Medical Treatment; Quality of Life Scores at 12 and 24 Months
Keywords: Intermittent claudication; Superficial femoral artery; Stenting; Medical treatment; Quality of life
MeSH Terms: conditions — Intermittent Claudication | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stenting (Active Comparator): Active treatment group
  Interventions: Procedure: Stenting
- Conservative treatment (Placebo Comparator): Best medical treatment
  Interventions: Other: Best medical treatment

INTERVENTIONS:
Procedure: Stenting — The stent should be deployed percutaneously, appropriate stent(s) size selected based upon the angiogram. The diameter must be 1-2 mm larger than the vessel. Length is chosen to cover lesion with one stent if possible. The choice of brand will be made through random selection among those offering possibility to cover the lesion with one stent. If more than one stent is required, overlap between 0.5 and 1 cm is acceptable. Postdilatation must be performed with a PTA balloon shorter than the length and less than the diameter of the stent. An angiogram should be made to compare the pre- and post-implant minimum lumen diameters. The non-diseased artery diameters shall be measured and residual % stenosis calculated.
  Other Names: Endovascular treatment of claudication
  Arms: Stenting
Other: Best medical treatment — Patients randomised to conservative treatment will receive appropriate medication with target levels of cholesterol 4,5 mmol/l, LDL 2,5 mmol/l and blood pressure level of 130/80 mmHg in addition to instruction how to engage in an exercise program. Each patient will receive a 'step-meter' which has to be carried during all activity during the first month and then during one week before each follow up visit. Step-meter read-outs will be recorded during each follow up visit. Smokers will be actively advised to quit smoking.
  Other Names: Medical treatment of intermittent claudication
  Arms: Conservative treatment

SUMMARY:
The aim of this study is to evaluate whether primary stenting with self expanding stent in patients with peripheral arterial disease suffering from stable claudication due to superficial femoral artery disease results in improved patient outcomes, compared to conservative treatment alone as measured by improvement in Quality of Life scores at 12 months after treatment using established surveys. Patients will be followed up 24 months after treatment. Planned recruitment and randomization of 100 patients was completed June 2015.

DETAILED DESCRIPTION:
Occlusive disease of the femoro-popliteal arteries is associated with symptoms ranging from pain in the calf on exertion to pain at rest and ultimately ulceration and gangrene. Treatment options include a) conservative measures, with attention to medical risk factors, smoking cessation and exercise programmes, b) minimally invasive treatments such as angioplasty and c) surgical procedures such as femoro-popliteal bypass grafts.

Percutaneous transluminal angioplasty (PTA) has been widely used in the treatment of femoro-popliteal stenosis and occlusion for many years. However, the medium and long-term results have always been suboptimal due to a high rate of restenosis.

With restenosis rates of 70 % with PTA alone in long SFA lesions. Factors which contribute to poor results include the presence of occlusion rather than stenosis, the length of the lesion and the severity of run-off vessel disease.(1)

Stents are expandable metal mesh tubes which are widely used in the treatment of arterial disease in the coronary, renal and iliac arteries, where they have been shown to have superior patency to balloon angioplasty alone.

In the treatment of SFA lesions several early studies have investigated the patency of balloon expandable stents. These are stents with low flexibility and high risk of deformation in SFA. Medium and long-term results are not better than with PTA alone.(2)

Self expanding nitinol stents are stents generally with high flexibility and moderate to high radial force. Initial studies have shown promising results in the SFA.(3)

Early prospective randomised studies , the Sirocco I and II study show as low as 7 % restenosis rate at 6 months and 18% at 12 months self expanding nitinol stent.(4, 5) Later studies have focused on the issue of the correlation of stent fractures and low patency. These have shown that higher restenosis rates correlated to the length of the stented segment, number of stents and stent brand (6)

Up to now the most frequent use of stents in the SFA is "bailout" stenting. Investigated in a prospective randomised trial on patients with severe claudication or critical ischemia with long lesions (130 +- 60 mm) primary stenting in the SFA is showing superior results to PTA with bailout stenting on restenosis rate, ABI and walking distance.(7) There are for the moment two more trials investigating the results of direct stenting.

The FAST trial investigated claudicants with short lesions (4,5 cm); the stent arm used Luminexx stents versus PTA alone with no significant in difference in patency between both treatment arms after 12 months follow up.(8) The Resilient trial investigated patients with claudication and critical limb ischemia with 6,5 cm long lesions. The results are not published, but positive "pre hand" information has already come out. (9)

The most accepted treatment in claudicants is conservative best medical treatment with or without supervised walking training.(10) There is a trend to stent treatment in certain situations.

There are to the best of our knowledge no studies comparing direct stenting with conservative treatment in claudicants.

The aim of this study is to evaluate whether primary stenting with nitinol self expanding stent in patients suffering from stable claudication (Fontaine IIa and IIb) due to superficial femoral artery disease, results in improved patient outcomes, compared to conservative treatment alone as measured by improvement in Quality of Life scores at 12 months after treatment using SF-36 and EuroQol EQ-5D surveys. Patients will be followed up 24 months after treatment.

A secondary objective is to study the impact of primary stenting versus conservative treatment on ABI and Walking Distance development during the 24 month follow up period. In addition, cost-parameters will be collected in each arm to allow for basic cost-effectiveness comparisons after 24 months.

12 month follow-up data have been published in Eur J Vasc Endovasc Surg 2017;53:686-694. All 24 month follow-up data have been collected, and a manuscript is in preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Female patients with child bearing potential may not be pregnant at study entry and must utilize reliable birth control for the duration of their participation in the study.
3. Patient suffering from stable claudication (Fontaine IIa and IIb).
4. One de-novo or restenotic superficial femoral artery with the target treatment area not extending beyond approximately 3 cm above the patella at MRA.
5. Patent popliteal artery on the index side, and runoff vessel situation at level six or better according to Rutherford classification prior to the day of the procedure. Target vessel diameter ≥ 4 mm at MRA.
6. Patient is willing and able to comply with the specified follow-up evaluation
7. The patient or legally authorized representative must provide written informed consent prior to the procedure.

Exclusion Criteria:

1. Recent hemorrhagic stroke (within past 3 months)
2. Aneurysm in the SFA or popliteal artery
3. Previously implanted stent(s) in the to be treated artery at the same site
4. Poor aortoiliac or common femoral "inflow", which would be deemed inadequate to support a femoropopliteal bypass graft. However, intervention to restore adequate blood flow at least three months prior to the index procedure is allowed
5. Significant vessel tortuosity or other parameters prohibiting access to the lesion or 90° tortuosity which would prevent delivery of the stent device
6. Revascularisation involving the same limb 30 days prior to the index procedure or a planned revascularisation within 30 days after the index procedure

8.Critical Limb Ischemia in the index leg (Fontaine III and IV). 9.Requirement of stent placement in the popliteal artery. For the purpose of this protocol all lesions are to be located at least three centimetres proximal to the superior edge of the patella.

10.Life expectancy of less than 24 months or other factors making clinical follow-up difficult 11.Patients enrolled in this or other clinical trial or anticipated to be included into a trial, without written approval of principal investigator of this study.

12.Walking capacity more than 500 meters.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Improvement in Quality of Life scores | 12 months
  Improvement in Quality of Life scores at 12 months after treatment using SF-36 and EuroQol EQ-5D surveys

SECONDARY OUTCOMES:
Ankle/Brachial Index (ABI) and Walking Distance | 24 months
  Ankle/Brachial Index (ABI) and walking distance development during the follow up period. In addition, cost-parameters will be collected in each arm to allow for basic cost-effectiveness comparisons after 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Lindgren, MD, Principal Investigator — Dept of Radiology, Helsingborg Hospital, Helsingborg, Sweden
Locations (2):
- Sweden (2):
  - Dept of Radiology, Helsingborg Hospital, Helsingborg
  - Department of Vascular Disease, Skåne University Hospital, Malmo

REFERENCES:
- [Result] Lindgren H, Qvarfordt P, Akesson M, Bergman S, Gottsater A; Swedish Endovascular Claudication Stenting Trialists. Primary Stenting of the Superficial Femoral Artery in Intermittent Claudication Improves Health Related Quality of Life, ABI and Walking Distance: 12 Month Results of a Controlled Randomised Multicentre Trial. Eur J Vasc Endovasc Surg. 2017 May;53(5):686-694. doi: 10.1016/j.ejvs.2017.01.026. Epub 2017 Mar 31. PMID 28372983
- [Derived] Lindgren HIV, Qvarfordt P, Bergman S, Gottsater A; Swedish Endovascular Claudication Stenting Trialists. Primary Stenting of the Superficial Femoral Artery in Patients with Intermittent Claudication Has Durable Effects on Health-Related Quality of Life at 24 Months: Results of a Randomized Controlled Trial. Cardiovasc Intervent Radiol. 2018 Jun;41(6):872-881. doi: 10.1007/s00270-018-1925-0. Epub 2018 Mar 8. PMID 29520431